CLINICAL TRIAL: NCT02439476
Title: Non-interventional Study Evaluating Plerixafor-based Mobilization for Salvage Autologous Hematopoietic Stem Cell Transplantation in Relapsed Myeloma
Brief Title: Non-interventional Study on Salvage Auto in Relapsed Myeloma
Acronym: IFM-2015-03
Status: Completed | Type: Observational
Sponsor: Association for Training, Education, and Research in Hematology, Immunology, and Transplantation (Other)
Responsible Party: Sponsor
Other Study IDs: IFM-2015-03
Record Dates: First submitted 2015-04-27; First posted 2015-05-08 (Estimated); Last update posted 2021-01-20 (Actual); Status verified 2020-05

CONDITIONS: Relapsed Multiple Myeloma
Keywords: Multiple myeloma; ASCT; plerixafor; stem cell mobilization; Salvage ASCT using plerixafor-based stem cell mobilization in relapsed multiple myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Relapsed multiple myeloma patients who are considered eligible: Patients mobilized using G-CSF+Plerixafor according to Plerixafor label in France will be included. Apheresis will be performed according to standard practice and local guidelines. Once the autologous stem cell product becomes available, patients will undergo ASCT conditioned by high dose Melphalan according to standard practice in each centre

SUMMARY:
Multiple myeloma (MM) is an incurable disease that is characterized by the accumulation of clonal plasma cells in the bone marrow. While MM patients with relapsed disease may achieve responses to subsequent antimyeloma therapies, the duration of response decreases with successive relapses until resistant disease develops. Until recently, the median survival following relapse after induction therapy was approximately one year. The relatively recent US Food and Drug Administration (FDA) approvals of bortezomib (2003) and combination lenalidomide plus dexamethasone (2006) therapies for the treatment of previously treated MM has provided effective therapeutic options that give patients with relapsed or refractory MM the prospect for a prolongation of overall and progression-free survival times. However, MM remains an incurable disease. A clear unmet medical need still exists for additional novel therapeutic options for the treatment of previously treated MM.

Plerixafor reversibly inhibits CXCR4 binding to stromal cell derived factor (SDF)-1alpha and was recently discovered to be an effective agent to mobilize CD34+ cells into the peripheral blood. In normal volunteers, administering Plerixafor after 4-5 days of G-CSF resulted in a 3-3.5 fold increase in circulating CD34+ cells. Two phases 3 studies demonstrated that the combination of G-CSF and Plerixafor is superior to G-CSF alone for mobilizing hematopoietic progenitor cells in front-line or as salvage therapy in patients with multiple myeloma.

Nevertheless, almost all patients ultimately relapse, and no plateau is observed in the survival curves. At the time of disease recurrence, there is not one standard salvage approach, but instead, various therapeutic options are available, including novel agents-based therapy, administered for a fixed duration of time or until progression. In the pivotal trial for the approval of bortezomib as monotherapy in relapsed and refractory MM, the median PFS was 7 months, whereas in the pivotal trials for the approval of lenalidomide in combination with dexamethasone in the same group of patients, the median time to progression was approximately 11 months. A more recent prospective, randomized, phase 3 study has shown that a triplet combination of bortezomib, thalidomide and dexamethasone (VTD) achieved superior results compared to thalidomide dexamethasone (TD) alone in patients relapsing following ASCT, with a median time to progression of 19.5 versus 13.8 months, respectively. This study suggests that combinations consisting of both an IMiD and a proteasome inhibitor are a valuable option at the time of relapse.

However, when a frozen graft is available, it is also possible to repeat high-dose therapy in patients who previously responded to the frontline application of high-dose melphalan and ASCT. Over time, several reports have demonstrated the feasibility of this salvage strategy. The majority of data are available from retrospective studies and are based on single-centre experiences with small numbers of selected patients. In this setting, PFS has been shown to range from 7 to 22 months, and the treatment-related mortality (TRM) was acceptable, ranging from 0 to 8%. Various prognostic factors for prolonged PFS have been described, such as the duration of response to the first high-dose therapy, or the number of lines of therapy prior to salvage ASCT.

With this background, this prospective non-interventional multicentre study will aim to collect data on the feasibility of salvage ASCT using a Plerixafor-based stem cell mobilization in relapsed MM, according to Plerixafor label in France.

This is a non-interventional study; visit will be performed as usual, according to each center practices. No additional visits will be requested for the study purpose. The date for each visit and any data generated must be recorded on the appropriate eCRF.

The study will consist of 3 periods:

* An early screening period
* Autologous stem cell mobilization period
* High dose melphalan therapy and autologous graft infusion and follow-up for12 months after salvage ASCT Inclusion visit

This visit may occur up to 28 days before Mozobil® administration. This visit will be performed during the visit of pre-transplant assessment. For the pre-transplant assessment, the procedures are performed routinely before ASCT even if the patient is not included in the study:

Stem cell mobilization phase The stem cell mobilization phase is performed according to standard practice of each participating centre.

Follow-up visits High dose melphalan administration and autologous graft infusion will be performed according to each centre standard practice. Patients will be followed according to each center practices. The follow-up of this non-interventional study will end 12 months after ASCT.

Subjects will be enrolled over a 2 years period. The total duration of the study will be 36 months

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥ 18 years,
* Relapsed myeloma according to standard criteria and eligible for a second salvage autologous transplantation. Eligibility to autologous transplantation is based on local guidelines and standard practice
* Written patient's agreement

Exclusion Criteria:

* Age > 75,
* Contraindication to autologous stem cell transplantation
* Contraindications to the use of plerixafor

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Relapsed multiple myeloma patients will be recruited in sites from the French collaborative IFM group in France
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2016-08-08 (Actual); Primary Completion 2020-08-08 (Actual); Study Completion 2020-08-08 (Actual)

PRIMARY OUTCOMES:
Feasibility to collect at least 2x10e6/kg CD34+ peripheral blood cell stem cells | from date of Plerixafor based mobilization until the date of stem cells transplantation, an expected average of 24 hours
  Percentage of patients achieving CD34+ ≥ 2x10e6/kg recipient body weight in one apheresis session after stem cell mobilization

SECONDARY OUTCOMES:
Engraftment after ASCT (neutrophil and platelets recovery) | Time to achieve neutrophil (>500/µl) and platelets (first of three days with>20G/l without transfusion), an expected average of 20 days
Time to disease progression | from the date of ASCT to the date of the first observation of disease progression, assessed up to 12 months follow-up
Duration of response | the time from partial response or complete response to the first documentation of disease progression, assessed up to 12 months follow-up
Progression free survival (PFS) | time from the start of treatment to the first documentation of disease progression or death from any cause during study, whichever occurs earlier, assessed up to 12 months follow-up
Overall Survival | from the date of ASCT to the date of death or the last date the patient was known to be alive whichever occurs first, assessed up to 12 months follow-up
Clinical Safety as measured by the type, the frequency and the severity of adverse events and laboratory abnormalities | 12 months follow-up
  incidence of treatment emergent Adverse event (TEAE), serious adverse event (SAE) and laboratory abnormalities using NCI common toxicity criteria

CONTACTS AND LOCATIONS:
Locations (1):
- Hématologie Clinique, Hôpital Saint Antoine, Paris, France

REFERENCES:
- [Derived] van de Wyngaert Z, Malard F, Hulin C, Caillot D, Mariette C, Facon T, Touzeau C, Perrot A, Moreau P, Hebraud B, Kanouni T, Heshmati F, Lebon D, Mohty M, Chabannon C. Non-interventional Study Evaluating the Mobilization of Stem Cells by Plerixafor Before Salvage Autologous Stem Cell Transplant in Relapsed Multiple Myeloma (IFM-2015-03). Clin Hematol Int. 2023 Mar;5(1):38-42. doi: 10.1007/s44228-023-00030-0. Epub 2023 Feb 12. PMID 36781774